CLINICAL TRIAL: NCT01537653
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability and Pharmacokinetics of Ascending Single Subcutaneous Doses of SAR231893/REGN668 in Healthy Japanese Adult Male Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of SAR231893 (REGN668) in Healthy Japanese Adult Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDU12265; U1111-1127-2719 (Other: UTN)
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2013-12-06 (Estimated); Status verified 2012-11

CONDITIONS: Healthy
MeSH Terms: interventions — dupilumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- SAR231893 (REGN668), Dose Level 4 (Experimental): Dose Level 4
  Interventions: Drug: SAR231893 (REGN668)
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- SAR231893 (REGN668), Dose Level 1 (Experimental): Dose Level 1
  Interventions: Drug: SAR231893 (REGN668)
- SAR231893 (REGN668), Dose Level 2 (Experimental): Dose Level 2
  Interventions: Drug: SAR231893 (REGN668)
- SAR231893 (REGN668), Dose Level 3 (Experimental): Dose Level 3
  Interventions: Drug: SAR231893 (REGN668)

INTERVENTIONS:
Drug: SAR231893 (REGN668) — Pharmaceutical form:Solution in a vial Route of administration: Subcutaneous injection
  Arms: SAR231893 (REGN668), Dose Level 1; SAR231893 (REGN668), Dose Level 2; SAR231893 (REGN668), Dose Level 3; SAR231893 (REGN668), Dose Level 4
Drug: placebo — Pharmaceutical form:Solution in a vial Route of administration: Subcutaneous injection
  Arms: Placebo

SUMMARY:
Primary Objective:

Assess the safety and tolerability of SAR231893 (REGN668) after ascending single subcutaneous (SC) doses in healthy Japanese adult male subjects

Secondary Objectives:

Assess the following parameters after ascending single SC doses in healthy Japanese adult male subjects

* The pharmacokinetics of SAR231893 (REGN668)
* The immunogenicity of SAR231893 (REGN668)
* Exploratory analyses of the pharmacodynamics of SAR231893 (REGN668)

DETAILED DESCRIPTION:
Total duration of the study period per subject is 11 weeks broken down as follows:

Screening period = 2 to 21 days Treatment period = 57 days, including 1 treatment day

ELIGIBILITY:
Inclusion criteria:

* Japanese adult male subjects, between 20 and 45 years of age, inclusive.
* Body weight between 50.0 and 95.0 kg, inclusive, body mass index between 18.0 and 28.0 kg/m2, inclusive.
* Certified as healthy by a comprehensive clinical assessment.
* Having given written informed consent prior to undertaking any study-related procedure.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastrointestinal, hepatic, renal, metabolic, hematological, neurological, osteomuscular, articular, psychiatric, systemic, ocular, or infectious disease, or signs of acute illness.
* Any subject who cannot prohibit intensive physical activity throughout the study duration.
* Positive result on any of the following tests: hepatitis B surface (HBs Ag) antigen, anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, human immunodeficiency virus (HIV) antigen and antibodies.
* Positive result on urine drug screen (amphetamines/methamphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, opiates).
* Serum alcohol level over the upper limit of normal range (ULN).
* Previous exposure to any therapeutic or investigational biological agent.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Number of subjects with standard safety assessments (adverse events, physical examinations, 12 lead ECGs, vital signs and laboratory tests) | Up to 57 days

SECONDARY OUTCOMES:
Pharmacokinetics: Serum concentrations of SAR231893 (REGN668) over time | Up to 57 days
Pharmacodynamics: Serum total Immunoglobulin E (IgE) and Thymus and activation regulated chemokine (TARC) over time | Up to 57 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392001, Toshima-Ku, Japan

REFERENCES:
- [Derived] Li Z, Radin A, Li M, Hamilton JD, Kajiwara M, Davis JD, Takahashi Y, Hasegawa S, Ming JE, DiCioccio AT, Li Y, Kovalenko P, Lu Q, Ortemann-Renon C, Ardeleanu M, Swanson BN. Pharmacokinetics, Pharmacodynamics, Safety, and Tolerability of Dupilumab in Healthy Adult Subjects. Clin Pharmacol Drug Dev. 2020 Aug;9(6):742-755. doi: 10.1002/cpdd.798. Epub 2020 Apr 29. PMID 32348036